CLINICAL TRIAL: NCT02253862
Title: Assessment of Single-dose Oral Tadalafil Pharmacokinetic Characteristics When Simultaneously Co-administered With Single-dose and Steady-state Tipranavir/Ritonavir 500 mg/200 mg to Healthy Male Volunteers
Brief Title: Pharmacokinetic of Tadalafil Co-administered With Tipranavir/Ritonavir to Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1182.83
Record Dates: First submitted 2014-09-30; First posted 2014-10-01 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2014-09

CONDITIONS: Healthy
MeSH Terms: interventions — Tadalafil; tipranavir; Ritonavir

ARMS (1):
- Sequential treatment (Experimental)
  Interventions: Drug: Tadalafil; Drug: Tipranavir; Drug: Ritonavir

INTERVENTIONS:
Drug: Tadalafil — administered days 1, 8 and 16
Drug: Tipranavir — administered days 8-18
Drug: Ritonavir — administered days 8-18

SUMMARY:
Study to assess the effects of single-dose and steady-state tipranavir/ritonavir 500 mg/200 mg on the single-dose pharmacokinetics of tadalafil 10 mg

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Healthy male subjects aged between 18 years and 55 years inclusive
3. Weighing at least 40 kg
4. Volunteers must be hospitalized on day of pharmacokinetic assessments for each regimen
5. Volunteers must be willing to complete all study-related activities
6. Each volunteer must have a valid social security regimen
7. Each volunteer must have acceptable medical history, physical examination and laboratory test
8. Volunteers with negative HIV serology

Exclusion Criteria:

1. History or presence of allergy to the study drugs or their components or drugs of their class, or a history of drug or other allergy that, in the opinion of the physician responsible, contraindicates their participation. (If heparin is used during pharmacokinetic (PK) sampling, subjects with a history of sensibility to heparin or heparin-induced thrombocytopenia should not be enrolled)
2. Any finding of the medical examination (including blood pressure, pulse rate, and electrocardiogram) deviating from normal and of clinical relevance
3. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunologic, haematological, oncological or hormonal disorders
4. Known elevated liver enzymes in past clinical trials with any compound (experimental or marketed)
5. Clinically relevant laboratory abnormalities and all abnormal laboratory values >Grade 1, based on the Division of AIDS Grading Scale
6. Subjects with a history of any illness or allergy that, in the opinion of the investigator, might confound the results of the study or pose additional risk in administering tipranavir, ritonavir or tadalafil to the subject
7. Volunteers who are using any form of organic nitrate, either regularly and/or intermittently (contraindication to use tadalafil)
8. Hypersensitivity to tadalafil, tipranavir, ritonavir or their excipients
9. Concurrent treatment with other experimental compounds
10. Inadequate venous access
11. Contraindications to tadalafil: Volunteers with mild or moderate hepatic impairment, Renal insufficiency or Cardiovascular disease (patients with a myocardial infarction within the last 90 days, unstable angina or angina occurring during sexual intercourse, patients with New York Heart Association Class 2 or greater heart failure in the last 6 months, patients with uncontrolled arrhythmias, hypotension (<90/50 mm Hg), or uncontrolled hypertension (>170/100 mm Hg), and patients with a stroke within the last 6 months)
12. Clinically unacceptable result at the screening physical examination
13. Use of investigational medications within 30 days before study entry
14. Patients hospitalized in a medical or social establishment, for any other reason than research
15. People deprived of judicial or administrative freedom.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2005-12; Primary Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) for Tadalafil | up to 72 hours after drug administration
Plasma Concentration (Cp12h) for Tadalafil | 12 hours after drug administration
Area Under Plasma Concentration-time Curve (AUC0-72h) for Tadalafil | up to 72 hours after drug administration
AUC0-∞ for Tadalafil | up to 72 hours after drug administration

SECONDARY OUTCOMES:
Cmax for Tipranavir and Ritonavir | up to 12 hours after drug administration
Cp12 for Tipranavir and Ritonavir | 12 hours after drug administration
AUC0-12hTipranavir and Ritonavir | 12 hours after drug administration
Time of Maximum Concentration | up to 72 hours after drug administration
Elimination half-life (t1/2) | up to 72 hours after drug administration
Total body clearance (Cl/F) | up to 72 hours after drug administration
Volume of distribution, | up to 72 hours after drug administration
Number of subjects with adverse events | up to 42 days